CLINICAL TRIAL: NCT03205033
Title: Melatonin as a Circadian Clock Regulator, Neuromodulator and Myelo-protector in Adjuvant Breast Cancer Chemotherapy: a Randomized, Double-blind, Placebo-controlled Trial.
Brief Title: Melatonin as a Circadian Clock Regulator, Neuromodulator and Myelo-protector in Adjuvant Breast Cancer Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-0701
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-01

CONDITIONS: Sleep Disorders, Circadian Rhythm; Depression; Genotoxicity; Pain
Keywords: Melatonin; Breast cancer; Chemotherapy; Sleep-wake rhytms; Circadian rhythms
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Depression; Pain; Breast Neoplasms | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Active Comparator): Melatonin 20 mg Oral Capsules, once a day at bedtime
  Interventions: Drug: Melatonin 20 MG Oral Capsule
- Placebo (Placebo Comparator): Placebo Oral Capsules, once a day at bedtime
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Melatonin 20 MG Oral Capsule — 1 capsule/day 1 hour before go to bed
  Other Names: MTN
  Arms: Melatonin
Drug: Placebo oral capsule — 1 capsule/day 1 hour before go to bed
  Other Names: PCB
  Arms: Placebo

SUMMARY:
Breast cancer is the second most common cancer in the world, the most common in women, representing the leading cause of death in Brazil. The therapeutic approach for breast cancer includes surgery, radiotherapy, chemotherapy and endocrine therapy. Chemotherapy courses with side effects because the cytotoxic effects affect indistinctly neoplastic cells and normal cells. The cancer per se may promote disruption in circadian rhythm. Chemotherapy induces or enhances desynchronization of the sleep-wake cycle, which competes with impaired memory, mood, pain and poor quality of life. Melatonin is an attractive therapeutic option in this context. This neurohormone also has immunomodulatory, co-analgesic and anti-depressant properties. Additionally, the antioxidant properties of melatonin may decrease free radical formation, reducing damage to DNA. The objective is to assess the response to melatonin as a synchronizer of the sleep-wake rhythm, neuromodulator, and mieloprotetor genoprotetor in the effects induced by chemotherapy in women with breast cancer.

DETAILED DESCRIPTION:
This is a randomized, double-blind clinical trial, parallel, placebo-controlled trial. Breast cancer women treated surgically and with indication for adjuvant chemotherapy, aged between 18 and 75 years will be included. Patients will be randomized to receive 20mg of melatonin or placebo at bedtime. Treatment will initiate seven days before the start of chemotherapy to three days after the first cycle, totaling ten days. The sleep-wake rhythm will be assessed by actigraphy, which use will precede three days to start treatment. We will also evaluate the sleep-wake cycle by sleep diary. Other parameters will be measured as depressive symptoms, pain threshold pressure, effect on platelets and white series, the pain response to conditioned stimuli and quality of life. Serum markers of neuroplasticity will be measured as the Derivate Nerve Factor Brain BDNF and S100 β. The icronucleus effect will quantified by cell material from the oral mucosa. We expect that the use of melatonin, as a competitor to chemotherapy and synchronizer, improves tolerance to adjuvant treatment of breast cancer chemotherapy adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosed with breast cancer
* Indicated for the adjuvant treatment for breast cancer
* Between 18 years and 75 years
* Alphabetized

Exclusion Criteria:

* Undergone chemotherapy or radiotherapy before inclusion in the study.
* Pregnant
* Epilepsy
* Brain Stroke
* Multiple sclerosis
* BMI above 45 kg / m 2

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the response to melatonin as a sleep-wake rhythm synchronizer on the effects induced by chemotherapy in women with breast cancer. | 1 capsule of melatonin 20 mg or Placebo capsule, once a day, 1 hour before go to bed
  Actigraphy to assess the circadian rhythm

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Palmer ACS, Souza A, Dos Santos VS, Cavalheiro JAC, Schuh F, Zucatto AE, Biazus JV, Torres ILDS, Fregni F, Caumo W. The Effects of Melatonin on the Descending Pain Inhibitory System and Neural Plasticity Markers in Breast Cancer Patients Receiving Chemotherapy: Randomized, Double-Blinded, Placebo-Controlled Trial. Front Pharmacol. 2019 Nov 22;10:1382. doi: 10.3389/fphar.2019.01382. eCollection 2019. PMID 31824318